CLINICAL TRIAL: NCT03727581
Title: Dialysis Catheter Insertion With Substernal Ultrasound Guidance
Brief Title: Ultrasound for Guidewire Detection
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Krzysztof Letachowicz, Principal Investigator, Wroclaw Medical University
Other Study IDs: st40
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Kidney Failure, Acute; Kidney Failure, Chronic
Keywords: hemodialysis; vascular access; dialysis catheter
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound guidance — Jugular vein is punctured with ultrasound guidance and guidewire is advanced. Right atrium and inferior vena cava junction is visualized by ultrasound using substernal view. Presence of guidewire in inferior vena cava or right atrium is confirmed. The procedure of catheter insertion is continued.

SUMMARY:
The aim of the project is to check if there is a possibility for a nephrologist to visualise the guidewire by means of available ultrasound scanners. To evaluate that, the procedure of catheter insertion will be expanded by ultrasound examination of right atrium and inferior vena cava border using substernal view. Such imaging seems to ameliorate the safety of catheter implementation and could be a good alternative for fluoroscopy, eliminating its adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Renal failure requiring hemodialysis through a dialysis catheter
* Capable of giving informed consent
* Placement of internal jugular vein catheter

Exclusion Criteria:

* Inability to provide informed consent
* Poor visualisation of inferior vena cava

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute kidney disease or end stage renal disease who need dialysis catheter insertion for hemodialysis performance
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Successful guidewire insertion | 5 minutes
  Visualization of guidewire in right atrium-inferior vena cava junction
Successful catheter placement | 2 hours
  Catheter tip in lower part of superior vena cava or right atrium on chest x-ray. Good catheter function.

SECONDARY OUTCOMES:
Complication rate | 24 hours
  Presence of pneumothorax, hematoma, catheter dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Letachowicz, MD, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Department of Nephrology and Transplantation Medicine, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No